CLINICAL TRIAL: NCT05123521
Title: Incidence of Drug Abuse at the Cairo University Teaching Hospital Among Patients Who Underwent Elective Surgeries
Brief Title: Drug Abuse Among Elective Surgeries: an Observational Study.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, associate prof, Cairo University
Other Study IDs: amera master
Record Dates: First submitted 2021-10-23; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Drug Abuse
Keywords: drug abuse; Cairo Teaching Hospital; elective surgery
MeSH Terms: conditions — Substance-Related Disorders | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: urine analysis — Urine was then tested for evidence of substance abuse using the multi-drug screen panel dip steak ABONtm (Abon Biopharm (Hangzhou) CO., Ltd) which is a lateral flow chromatographic immunoassay . It allowed for qualitative detection of multiple drugs in a single run. This kit was chosen for its ability to detect the most commonly abused substances in Egypt, namely: opioids, benzodiazepines, hashish, and tramadol. A single coloured line at region C for of a specific drug indicated a positive result, whilst two coloured lines at both regions C and T indicated a negative result. The absence of coloured lines was an indication of the invalidity of the particular kit, and the kit was discarded.

SUMMARY:
Drug abusers and addicts form a challenge to the anesthetist because of the added potential risks involved in the administration of anesthesia to this subset of patients, including potential unforeseen drug-drug interactions. In this study, we aimed at screening all patients scheduled for elective orthopedic or general surgeries at the Cairo University Teaching Hospital during a set period of time for the most commonly abused drugs in Egypt.

DETAILED DESCRIPTION:
All patients included in the study consented to take part in this study. Each patient was asked to answer a questionnaire and submit a urine sample in order to be screened for the most commonly abused drugs in Egypt (hashish, tramadol, benzodiazepine, and morphine). Patients were then followed up both intra and post-operatively. Values of patient vital signs, Richmond Agitation-Sedation Scale (RASS) scores as well as clinical recovery scores (CRS) were all diligently recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients classified as American Society of Anaesthesiology (ASA) I or II patients
* patients between 15 and 60 years of age
* patients scheduled for elective surgery.

Exclusion Criteria:

* emergency surgery
* those with disturbed conscious levels
* history of psychological illness
* who refused to give consent

Ages: 15 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: those who had presented to the General Surgery or Orthopaedics Departments
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
urine analysis | THREE MONTHS
  multi-drug screen panel dip steak (Abon Biopharm (Hangzhou) , Ltd)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Ali, Md, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No